CLINICAL TRIAL: NCT00981318
Title: Pilot Assessment of Lopinavir/Ritonavir and Maraviroc in Experienced Patients
Brief Title: Pilot Assessment of Lopinavir/Ritonavir and Maraviroc
Acronym: PALM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to enroll expected number of subjects
Sponsor: Rodwick, Barry M., M.D. (Individual)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Barry M. Rodwick, M. D., Principal Investigator, Rodwick, Barry M., M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rodwick01
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: Acquired Immunodeficiency Syndrome; HIV; AIDS; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; Maraviroc; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lopinavir/ritonavir 400/100 mg bid plus maraviroc 150 mg bid (Other): single arm
  Interventions: Drug: lopinavir/ritonavir plus maraviroc

INTERVENTIONS:
Drug: lopinavir/ritonavir plus maraviroc — lopinavir/ritonavir 400/100 mg bid plus maraviroc 150 mg bid
  Other Names: Kaletra; lopinavir; Selzentry

SUMMARY:
This is a study to assess the response of lopinavir/ritonavir plus maraviroc (with no nucleoside medications) in HIV patients failing their initial antiviral therapy.

DETAILED DESCRIPTION:
As long-term toxicity to many of the nucleoside medications have become known, interest has increased in treatment regimens that do not use these medications. This study is to assess the response of one such "nucleoside-sparing" therapy in patients who are showing failure to their initial nucleoside-containing treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV viral load > 1,000 on current antiviral medications
* No resistance to study medications
* Over 18 years of age

Exclusion Criteria:

* Hepatitis B co-infection
* Pregnancy
* Previous therapy with either of the study medications
* Ongoing substance abuse
* Significant history of other physical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Virologic response defined as viral load reduction of >/= 1 log | 48 weeks

SECONDARY OUTCOMES:
Assess proportion of patients with HIV-1 viral load < 48 copies | 48 weks
Assess time to loss of virologic response | 48 weeks
Assess development of resistance mutations in patients who develop rebound | 48 weeks
Compare serum lipid profile changes | 48 weeks
Assess safety and tolerability | 48 weeks
Assess degree of immune reconstitution | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry M. Rodwick, M. D., Principal Investigator — Barry M. Rodwick, M. D.
Locations (1):
- Barry M. Rodwick, M. D., Safety Harbor, Florida, United States